CLINICAL TRIAL: NCT05914051
Title: PRELOAD TAVI Trial: Prospective Randomized Trial of Volume Preload Optimization in Patients With Severe Aortic Stenosis Treated on Spontaneous Breathing With Transfemoral TAVI
Brief Title: PRELOAD-TAVI Trial
Acronym: PRELOAD-TAVI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación de investigación HM (Other)
Responsible Party: Principal Investigator, Leire Unzue Vallejo, PRELOAD-TAVI Trial, Fundación de investigación HM
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRELOAD-TAVI
Record Dates: First submitted 2023-03-23; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: TAVI

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Volume preload optimization. (Experimental): Volume overload with 250 cc saline solution will be performed in the intervention arm, verifying the response of the cardiac output and stroke volume with non invasive continue monitoring.
  Interventions: Other: Colloid preload
- Control group (No Intervention): Standard care without volume preload.

INTERVENTIONS:
Other: Colloid preload — 250 cc of colloid preload solution will be infused in the intervention group
  Arms: Volume preload optimization.

SUMMARY:
The aim is to assess the response of cardiac output and stroke volume to volume preload optimization in patients with severe aortic stenosis treated with aortic prosthesis implantation.

DETAILED DESCRIPTION:
Patients with severe aortic stenosis present a maintained overload pressure of the left ventricle that can lead to a progressive hypertrophy. This results in elevated left-sided filling pressures and impaired diastolic function.In this context, paradoxical changes in left ventricular function after aortic valve replacement have been described, with acute decrease of the afterload condition that can result in the development of a dynamic intraventricular gradient, especially in the presence of small ventricles with severe hypertrophy, resulting in hemodynamic collapse.

In this setting, it is particularly important to ensure accurate left ventricular preload to optimize myocardial contractility and guarantee an adequate hemodynamic response to valve implantation.

Patients with severe aortic stenosis submitted for transfemoral TAVI on spontaneous breathing will be randomly assigned 1:1 to standard care vs volume preload optimization. Non-invasive continuous monitoring (Clear Sight System, Edwards Lifesciences) will be used to evaluate the cardiac output and the stroke volume in both groups, comparing the hemodynamics before and after valve implant.

ELIGIBILITY:
Inclusion Criteria:

* Aortic valve stenosis with echocardiographic derived criteria: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s or an initial aortic valve area of < 0.8 cm2

Exclusion Criteria:

* Cardiogenic shock.
* Life expectancy < 1 year.
* Need of mechanic ventilation.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac output after valve implant | "1 year"
  Cardiac output (l/min) after TAVI

SECONDARY OUTCOMES:
Stroke volume after valve implant | "1 year"
  SV (ml) after TAVI

OTHER OUTCOMES:
Need of inotropes | "1 year"
  Yes/no
HR after TAVI | "1 year"
  rpm

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: At recruitment and after study conclusion